CLINICAL TRIAL: NCT01947933
Title: A Phase I, Randomized, Placebo-Controlled Study of LY3074828, an Anti-IL-23 Humanized Antibody
Brief Title: A Safety Study of Mirikizumab (LY3074828)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15039; I6T-MC-AMAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-02

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — mirikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo IV (Placebo Comparator): Participants with psoriasis will receive a single dose of placebo matching mirikizumab intravenously (IV)
  Interventions: Biological: Placebo - IV
- Mirikizumab IV (Experimental): Participants with psoriasis will receive a single escalating dose of 5 milligram (mg), 20 mg, 60 mg, 120 mg, 200 mg, 350 mg, or 600 mg mirikizumab, IV
  Interventions: Biological: Mirikizumab- IV
- Mirikizumab SC (Experimental): Healthy participants will receive a single dose of 120 mg mirikizumab subcutaneously (SC).
  Interventions: Biological: Mirikizumab - SC

INTERVENTIONS:
Biological: Mirikizumab- IV — Administered IV
  Other Names: LY3074828
  Arms: Mirikizumab IV
Biological: Mirikizumab - SC — Administered SC
  Other Names: LY3074828
  Arms: Mirikizumab SC
Biological: Placebo - IV — Administered IV
  Arms: Placebo IV

SUMMARY:
The main purpose of this study is to evaluate the safety of the study drug known as mirikizumab. The study will investigate how the body processes the study drug and how the drug affects the body. The study will last about 3 months for each participant.

ELIGIBILITY:
Inclusion Criteria (Psoriasis participants):

* Chronic plaque psoriasis based on an investigator confirmed diagnosis of chronic psoriasis vulgaris for at least 6 months prior to baseline
* Plaque psoriasis involving >2% body surface area (BSA) in affected skin other than the face and scalp at screening and baseline
* Are willing and able to washout topicals for at least 14 days before baseline on the 2 target lesions

Inclusion Criteria (Healthy participants):

* Are overtly healthy males or females, as determined by medical history and physical examination
* Are women not of childbearing potential
* Are between the ages of 18 and 65 years, inclusive, at the time of screening
* Have a body mass index between 18.5 and 32.0 kilogram per square meter (kg/m2), inclusive, and a minimum body weight of 55 kg
* Have clinical laboratory test results within normal reference range for the central laboratory, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the ERB governing the site

Exclusion Criteria (Psoriasis and healthy participants):

* Have received treatment with biologic therapies for psoriasis (such as monoclonal antibodies, including marketed or investigational biologic therapy). Prior or current use of biologics for indications other than psoriasis may be allowed with sponsor approval
* Within 28 days prior to baseline: have received systemic nonbiologic psoriasis therapy
* Within 14 days prior to baseline: have received topical psoriasis treatment
* Have presence of significant uncontrolled cerebro-cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, neurologic or neuropsychiatric disorders or abnormal laboratory values at screening that, in the opinion of the investigator, pose an unacceptable risk to the subject if participating in the study or of interfering with the interpretation of data
* Have had clinically significant symptomatic herpes zoster within 3 months of screening
* Show evidence of active or latent tuberculosis (TB)
* Have received live vaccine(s) (included attenuated live vaccines) within 1 month of screening or intend to during the study
* Have significant allergies to humanized monoclonal antibodies or any components of the mirikizumab product formulation or have a history of significant atopy
* Have had lymphoma, leukemia, or any malignancy within the past 5 years, except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years and cervical carcinoma in situ, with no evidence of recurrence within 5 years prior to baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST, Study Director — Eli Lilly and Company
Locations (2):
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterloo, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo, single dose, administered intravenously (IV)
- 5 mg LY3074828: 5 milligram (mg) LY3074828, single dose, administered IV
- 20 mg LY3074828: 20 mg LY3074828, single dose, administered IV
- 60 mg LY3074828: 60 mg LY3074828, single dose, administered IV
- 120 mg LY3074828: 120 mg LY3074828, single dose, administered IV
- 120 mg LY3074828 SC: 120 mg LY3074828, single dose, administered subcutaneously (SC)
- 200 mg LY3074828: 200 mg LY3074828, single dose, administered IV
- 350 mg LY3074828: 350 mg LY3074828, single dose, administered IV
- 600 mg LY3074828: 600 mg LY3074828, single dose, administered IV
Period: Overall Study
Arm/Group | Placebo | 5 mg LY3074828 | 20 mg LY3074828 | 60 mg LY3074828 | 120 mg LY3074828 | 120 mg LY3074828 SC | 200 mg LY3074828 | 350 mg LY3074828 | 600 mg LY3074828
Started | 7 | 3 | 5 | 5 | 5 | 5 | 5 | 5 | 5
Completed | 7 | 3 | 4 | 5 | 5 | 5 | 5 | 5 | 4
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: all randomized participants who received any amount of study drug.
Groups:
- Placebo: Placebo administered intravenously (IV)
- 5 mg LY3074828: 5 mg LY3074828 administered IV
- 20 mg LY3074828: 20 mg LY3074828 administered IV
- 60 mg LY3074828: 60 mg LY3074828 administered IV
- 120 mg LY3074828: 120 mg LY3074828 administered IV
- 120 mg LY3074828 SC: 120 mg LY3074828 administered subcutaneously (SC)
- 200 mg LY3074828: 200 mg LY3074828 administered IV
- 350 mg LY3074828: 350 mg LY3074828 administered IV
- 600 mg LY3074828: 600 mg LY3074828 administered IV
- Total: Total of all reporting groups
Arm/Group | Placebo | 5 mg LY3074828 | 20 mg LY3074828 | 60 mg LY3074828 | 120 mg LY3074828 | 120 mg LY3074828 SC | 200 mg LY3074828 | 350 mg LY3074828 | 600 mg LY3074828 | Total
Number analyzed (Participants) | 7 | 3 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.7 (13.39) | 51.0 (13.08) | 43.4 (13.32) | 44.0 (9.14) | 43.8 (13.33) | 37.2 (13.33) | 53.2 (14.55) | 37.4 (11.37) | 42.2 (10.57) | 43.8 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 4 | 0 | 2 | 5 | 2 | 1 | 2 | 18
  Male | 7 | 1 | 1 | 5 | 3 | 0 | 3 | 4 | 3 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 7 | 3 | 5 | 5 | 5 | 4 | 5 | 5 | 5 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 7 | 3 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  Canada | 7 | 3 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Adverse Event(s) (AEs) Considered by the Investigator to Be Related to Study Drug Administration
Description: This outcome has the list of adverse events which are related to the study drug. A summary of AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline through Week 12
Population: Safety Population: all randomized participants who received any amount of study drug.
Measure: Number; unit: Participants
Groups:
- 5 mg LY3074828: 5 mg LY3074828, single dose, administered IV
Arm/Group | Placebo | 5 mg LY3074828 | 20 mg LY3074828 | 60 mg LY3074828 | 120 mg LY3074828 | 120 mg LY3074828 SC | 200 mg LY3074828 | 350 mg LY3074828 | 600 mg LY3074828
Number analyzed (Participants) | 7 | 3 | 5 | 5 | 5 | 5 | 5 | 5 | 5
Participants | 1 | 1 | 2 | 0 | 0 | 3 | 1 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of LY3074828
Time Frame: IV Arms: Day 1 Predose, Postdose (End of Infusion, 2, 6 and 24h), Days 4, 8, 15, 22, 29, 43, 57, 71, and 85. SC Arm: Day 1 Predose, Postdose (6 and 24h), Days 4, 8, 11, 15, 22, 29, 43, 57, 71, and 85
Population: All randomized participants who received any amount of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg•day/mL (microgram•day/milliliters)
Groups:
- 120 mg LY3074828 SC: 120 mg LY3074828, single dose, administered SC
Arm/Group | 5 mg LY3074828 | 20 mg LY3074828 | 60 mg LY3074828 | 120 mg LY3074828 | 120 mg LY3074828 SC | 200 mg LY3074828 | 350 mg LY3074828 | 600 mg LY3074828
Number analyzed (Participants) | 2 | 5 | 5 | 5 | 5 | 5 | 5 | 5
μg•day/mL (microgram•day/milliliters) | NA (NA) — One participant not included in calculation of summary statistics. Geometric Mean and %CV not calculated for 2 participants. Values = Min 6.72, Max 8.40 | 33.6 (17) | 117 (15) | 287 (29) | 114 (49) | 366 (12) | 556 (25) | 1360 (23)

3. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3074828
Time Frame: as for outcome 2
Population: All randomized participants who received any amount of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL (microgram/milliliter)
Arm/Group | 5 mg LY3074828 | 20 mg LY3074828 | 60 mg LY3074828 | 120 mg LY3074828 | 120 mg LY3074828 SC | 200 mg LY3074828 | 350 mg LY3074828 | 600 mg LY3074828
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 5 | 5 | 5 | 5
μg/mL (microgram/milliliter) | 1.60 (22) | 5.34 (6) | 20.6 (29) | 41.1 (15) | 7.28 (23) | 68.8 (19) | 91.8 (6) | 220 (24)

ADVERSE EVENTS:
Arm/Group | Placebo | 5 mg LY3074828 | 20 mg LY3074828 | 60 mg LY3074828 | 120 mg LY3074828 | 120 mg LY3074828 SC | 200 mg LY3074828 | 350 mg LY3074828 | 600 mg LY3074828
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 6/7 | 3/3 | 5/5 | 5/5 | 2/5 | 4/5 | 4/5 | 4/5 | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=7) | 5 mg LY3074828 (N=3) | 20 mg LY3074828 (N=5) | 60 mg LY3074828 (N=5) | 120 mg LY3074828 (N=5) | 120 mg LY3074828 SC (N=5) | 200 mg LY3074828 (N=5) | 350 mg LY3074828 (N=5) | 600 mg LY3074828 (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 4 (4) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electric shock (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness exertional (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 0 (0) | 3 (3)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/2 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days